CLINICAL TRIAL: NCT07091006
Title: A Prospective Study on the Efficacy and Safety of Venetoclax, Azacitidine, and Homoharringtonine (VAH) Combination as a Bridging Regimen to Allogeneic Hematopoietic Stem Cell Transplantation in Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Efficacy and Safety of VAH as a Bridging Regimen to Allo-HCT in Relapsed/Refractory AML
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJ-BMT-013
Record Dates: First submitted 2025-07-07; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Relapse Leukemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Patients with relapsed/refractory acute myeloid leukaemia eligible for enrolment should be bridged with venetoclax, azacitidine, in combination with homoharringtonine before allo-HCT.
  Interventions: Drug: VAH

INTERVENTIONS:
Drug: VAH — For R/R AML patients, VAH bridging to conditioning regimen for allo-HCT.

SUMMARY:
Allogeneic hematopoietic cell transplantation (allo-HCT) is the only treatment that offers a possible cure for relapsed/refractory AML. Currently, the optimal preallo-HCT bridging regimen for relapsed/refractory AML patients is unclear. Venetoclax-based regimens, including Venetoclax + demethylating agents (HMA) , Venetoclax + HMA + other drugs and Venetoclax-based multidrug combinations as a bridging regimen improves response rate and post-transplant survival in relapsed/refractory AML patients. Therefore, the investigators conduct a prospective single-centre clinical study to evaluate the efficacy and safety of VAH as a transplant bridging regimen for relapsed/refractory AML.

DETAILED DESCRIPTION:
Relapsed/refractory acute myeloid leukaemia has an extremely poor prognosis, and allogeneic haematopoietic stem cell transplantation is the only treatment that offers the possibility of a cure for relapsed/refractory AML. Currently, the optimal pre-allo-HCT bridging regimen for relapsed/refractory AML patients is unclear. Previous studies have found that venetoclax and Azacitidine combined with homoharringtonine (VAH) bridging allogeneic transplantation for relapsed/refractory AML has a post-transplantation CRc of 78% and a 1-year OS of 85%, which is superior to other bridging regimens, and we have also found that VAH has a better safety and efficacy as a pre-transplantation bridging in our previous study. Therefore, the investigators propose to conduct a prospective single-centre clinical study to evaluate the efficacy and safety of VAH as a bridging regimen for transplantation in relapsed/refractory AML.

The aim of the study is assessment of the efficacy and safety of allogeneic haematopoietic stem cell transplantation for relapsed/refractory acute myeloid leukaemia in combination with venetoclax and Azacitidine in combination with homoharringtonine.

ELIGIBILITY:
Inclusion Criteria:

* Aged 14 to 70 years (inclusive), regardless of gender;
* The diagnosis of AML was confirmed on the basis of bone marrow cytomorphology, immunophenotyping and chromosomal and molecular biology tests;
* Relapsed AML: After achieving complete remission (CR), the reappearance of leukemic cells in peripheral blood, or ≥5% blasts in bone marrow (excluding other causes such as bone marrow regeneration after consolidation chemotherapy), or extramedullary infiltration by leukemic cells.

Refractory AML: Newly diagnosed cases that are unresponsive after two courses of standard induction therapy; patients who relapse within 12 months after consolidation/intensification therapy post-CR; patients who relapse after 12 months but fail to respond to conventional chemotherapy; patients with two or more relapses; or those with persistent extramedullary leukemia.

* With RUNX1::RUNX1T1 AML: Positive measurable residual disease (MRD) on bone marrow flow evaluation after the second consolidation therapy and/or less than a 3-log decrease in the RUNX1::RUNX1T1 fusion gene and diagnostic baseline values;
* ECOG score ≤2; HCT-CI score <3; Aspartate aminotransferase (AST) ≤ 3 times ULN (upper limit of normal, ULN); Alanine aminotransferase (ALT) ≤ 3x ULN; Total serum bilirubin ≤ 1.5 times the upper limit of normal ULN unless the patient has documented Gilbert syndrome; patients with Gilbert-Meulengracht syndrome with bilirubin ≤ 3.0 times the upper limit of normal and direct bilirubin ≤ 1.5 times the upper limit of normal may be included; Serum creatinine ≤ 1.5 times ULN or creatinine clearance ≥ 60 mL/min; Coagulation function: International Normalised Ratio (INR) ≤ 1.5 x ULN, Activated Partial Thromboplastin Time (APTT) ≤ 1.5 x ULN;
* Left ventricular ejection fraction (LVEF) ≥50%;

Exclusion Criteria:

* Allergies or contraindications to any of the drugs in the protocol;
* Currently have clinically significant active cardiovascular disease such as uncontrolled arrhythmias, uncontrolled hypertension, congestive heart failure, any grade 3 or 4 heart disease as determined by the New York Heart Association (NYHA) functional class, or a history of myocardial infarction within the 6 months prior to screening;
* Serious medical conditions that may limit the patient's participation in this trial (e.g., progressive infection, uncontrolled diabetes);
* Active autoimmune diseases such as SLE, rheumatoid arthritis, etc;
* Patients with neurological or psychiatric disorders;
* The patient is pregnant or breastfeeding;
* Those who are unable to understand or comply with the study protocol or are unable to sign the informed consent form.
* Other conditions that, in the opinion of the investigator, make the patient otherwise unsuitable for participation in this study;

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
2-year post-transplant relapse rate | through study completion, an average of 2 year
  relapse

SECONDARY OUTCOMES:
2-year event-free survival after transplantation | through study completion, an average of 2 year
  MRD positivity, relapse, death
Overall survival at 2 years after transplantation | through study completion, an average of 2 year
  survival

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoxia HU, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China